CLINICAL TRIAL: NCT04491370
Title: Safety and Tolerability of Myeloablative Conditioning and Autologous Stem Cell Transplantation Followed by Polatuzumab Vedotin (PV) Immunoconjugate Therapy in Patients With B-cell Non-Hodgkin and Hodgkin Lymphoma
Brief Title: Autologous Stem Cell Transplant Followed by Polatuzumab Vedotin in Patients With B-cell Non-Hodgkin and Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14357
Record Dates: First submitted 2020-07-16; First posted 2020-07-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: B-cell Lymphoma; Burkitt Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Transformed Non-Hodgkin Lymphoma; Richter Syndrome; Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Hodgkin Disease | interventions — polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Polatuzumab vedotin (Experimental): Evaluable patients for safety Patients receiving 1 dose of Polatuzumab Vedotin will be evaluable for safety.
  Evaluable patients for response Only in patients who are in PR or SD prior to PV and received a minimum of 3 doses will be evaluable.
  Evaluable patients for EFS, PFS, OS All patients who have completed conditioning and autoSCT will be evaluable for EFS, PFS, and OS.
  Interventions: Drug: Polatuzumab vedotin

INTERVENTIONS:
Drug: Polatuzumab vedotin — All patients will receive a myeloablative conditioning regimens (BEAM or CBV, as selected by the treating physician) followed by autologous stem cell transplant (ASCT). All patients on this study will receive an autologous stem cell transplant (ASCT) on Day 0 followed by supportive care including the drugs sargarmostim and filgrastim until blood counts are stable. If a complete, partial, or stable response is achieved following ASCT, the patient will receive an IV dose of Polatuzumab Vedotin once every 21 days until he/she receives 8 doses.

SUMMARY:
Patients will receive one of two conditioning regimens (BEAM or CBV) before receiving an autologous stem cell transplant (ASCT). If patients achieve either complete, partial, or stable response following ASCT, they will receive an IV dose of Polatuzumab Vedotin once every 21 days until they receive 8 doses. After Polatuzumab Vedotin therapy is completed, patients will be followed every 4 months for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis B-cell NHL: Burkitt lymphoma, Diffuse Large B Cell Lymphoma, Follicular Lymphoma, Mantle Cell Lymphoma, Marginal Zone Lymphoma, Transformed Follicular Lymphoma, Richter syndrome, and CD20+ Hodgkin Lymphoma.
* Disease Status Primary Induction Failure, 1st, 2nd or 3rd relapse/progression having attained a CR, PR, or stable disease post reinduction therapy.
* Performance Level Patients must have a performance status ≥ 50%. Use Karnofsky for patients > 16 years of age and Lansky for patients less than or equal to 16 years of age. See Appendix I for performance score.
* Life Expectancy Patients must have a life expectancy of > 6 weeks.
* Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study (4 weeks if prior nitrosourea).
  2. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent.
* Organ Function Requirements

Adequate Renal Function Defined As:

* Creatinine clearance or radioisotope GFR > 60 mL/min/1.73 m2 or
* A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female

* 12 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4
* 16 years 1.7 1.4

  * Adequate Liver Function Defined As:

    * Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) for age, and
    * SGOT (AST) or SGPT (ALT) < 3 x upper limit of normal (ULN) for age for presumed hepatic leukemia or lymphoma.
  * Adequate Cardiac Function Defined As:

    * Shortening fraction of > 27% by echocardiogram, or
    * Ejection fraction of > 50% by radionuclide angiogram.
  * Adequate Pulmonary Function Defined As:

    • Normal respiratory rate for age and a pulse oximetry > 94% on room air unless due to underlying malignancy.
  * Peripheral Blood Stem Cell Collection

    • Patients have a target of 5.0 x 106 CD34 (minimum of 2.5 x 106 CD34) PBSC collected and cryopreserved prior to start of myeloablative conditioning
  * All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

* Patient may not have had a prior stem cell transplant
* Patients must not have active CNS lymphoma
* Other concurrent investigational agents for treatment of B-cell lymphoma
* Pregnancy and/or active Breast Feeding
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation.
* Patient must not have an uncontrolled infection.
* Patient must not have ≥ Grade 3 neuropathy.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year
  To evaluate the safety and tolerability of Polatuzumab vedotin (PV) immunoconjugate therapy post myeloablative conditioning (MAC) and autologous stem cell transplantation (AutoSCT) in patients with B-cell non-Hodgkin lymphoma (NHL).
  Patients receiving 1 dose of Polatuzumab Vedotin will be evaluable for safety. To determine the safety events: Number of participants with treatment-related Grade III or higher adverse events as assessed by CTCAE v5.0.
  To determine the occurrence of any Grade ≥ 3 non hematologic toxicity (per CTCAE v.5) which is possibly, probably, or definitely related to polatuzumab vedotin.

SECONDARY OUTCOMES:
EFS, PFS, and OS | 2 years
  To measure event free survival (EFS), progression free survival (PFS) and overall survival (OS) in patients with B-cell NHL following MAC and AutoSCT and post AutoSCT PV maintenance therapy.
  All patients who have completed conditioning and autoSCT will be evaluable for EFS, PFS, and OS. EFS, PFS and OS will utilize Kaplan Meier product limit curve method. Response will be defined for patients with non-Hodgkin's lymphoma who had either measurable or detectable disease at the time of study entry in accordance with the revised IPNHL response criteria (Appendix VI) for patients ≤ 21 years of age and with the Lugano classification (Appendix VII) for patients > 21 years of age.
ORR | 2 years
  To measure overall response rate (ORR) of PV in B-cell NHL patients who are in PR or SD post MAC AutoSCT.
  Only in patients who are in PR or SD prior to PV and received a minimum of 3 doses will be evaluable. EFS, PFS and OS will utilize Kaplan Meier product limit curve method. Response will be defined for patients with non-Hodgkin's lymphoma who had either measurable or detectable disease at the time of study entry in accordance with the revised IPNHL response criteria (Appendix VI,[24]) for patients ≤ 21 years of age and with the Lugano classification (Appendix VII, [25]) for patients > 21 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Aliza Gardenswartz, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical Center, Valhalla, New York, United States